CLINICAL TRIAL: NCT02297022
Title: Phase 1 Study of Deep Brain Stimulation for the Treatment of Obesity in Patients With Prader-Willi Syndrome
Brief Title: Deep Brain Stimulation for the Treatment of Obesity in Patients With Prader-Willi Syndrome
Acronym: DBSPW
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InternalFunds
Record Dates: First submitted 2014-10-30; First posted 2014-11-21 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2014-11

CONDITIONS: Prader-Willi Syndrome
Keywords: Deep Brain Stimulation; obesity; Prader-Willi syndrome
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Patients with Prader-Willi syndrome to receive DBS.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation hypothalamic surgery in patients with Prader-Willi syndrome

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of deep brain stimulation in obese patients with Prader Willi syndrome refractory to conventional treatment.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and efficacy of deep brain stimulation in obese patients with Prader Willi syndrome refractory to conventional treatment. Patients will be implanted with hypothalamic DBS electrodes. Calorimetric and anthropometric measures, body mass index, side effects, neuropsychiatric evaluations will be carried out at 6 months for measuring primary and secondary outcome. Side effects will be monitored at 1, 3, 6 and 12 months following surgery.

ELIGIBILITY:
Inclusion Criteria:

* 15 years or older
* Parents able to give informed consent
* Diagnosis of Prader-Willi syndrome confirmed by genetic analysis
* Refractoriness to medical treatment, defined as a weight loss lower than 10% of the body weight with nutritional, pharmacological or surgical interventions
* Severe or morbid obesity
* No contra-indications to the surgical procedure

Exclusion Criteria:

* Cardiovascular disease that might significantly increase the surgical risk
* Brain lesions detected clinically or during MRI
* Use of cardiac pacemakers/ defibrillators
* Clinical conditions that may require the use of MRI in the post-operative period
* Patients undergoing chemotherapy or immunosuppressive treatments
* Patients unable to return to the hospital at the required intervals
* Previous neurosurgical treatments that may increase the risk of DBS surgery
* Active medical conditions that may require in-hospital treatment in the nearby future
* Previous diagnosis of epilepsy or status epilepticus
* Chronic infection
* Plan to use diathermy
* Metallic implants that might preclude MRI imaging of the brain
* Active participation in other experimental studies

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
waist circumference; mid-upper arm circumference | 6 months
resting energy expenditure | 6 months
Body mass index | 6 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 months

SECONDARY OUTCOMES:
daily food ingestion diary listing | 6 months
Child Yale-Brown Obsessive Compulsive Scale | 6 months
Child Behaviour Checklist | 6 months
Feeding Behaviour Questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Durval Damiani, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- HCFUMSP, São Paulo, São Paulo, Brazil